CLINICAL TRIAL: NCT01129713
Title: Comparison of Nexium Versus Secretol in the Healing and Controlling of Symptoms in Gastroesophageal Reflux Disease(GERD)Patients With Severe Erosive Esophagitis(EE).
Brief Title: Comparison of Nexium Versus Secretol in the Healing and Controlling of Symptoms in GERD Patients With Severe EE.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Effexus Pharmaceutical (Industry)
Collaborators: Southern Arizona VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEXIUM versus SECRETOL
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Heartburn; Indigestion
Keywords: GERD; Acid Reflux; Heartburn; Regurgitation; Indigestion
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Dyspepsia | interventions — Lansoprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nexium (Active Comparator): Comparing 40 mg.once daily in healing erosive esophagitis.
  Interventions: Drug: Nexium
- Secretol (Active Comparator): Comparing the efficacy of 80/80 Secretol once daily in healing erosive esophagitis.
  Interventions: Drug: Secretol

INTERVENTIONS:
Drug: Secretol — Comparing 80/80 once daily to Nexium once daily in healing erosive esophagitis.
  Other Names: lansoprazole/omeprazole combination
  Arms: Secretol
Drug: Nexium — Comparing 40 mg Nexium once daily to 80/80 Secretol once daily in healing erosive esophagitis.
  Other Names: Esomeprazole
  Arms: Nexium

SUMMARY:
To compare the complete healing of erosive esophagitis(EE) after 3 weeks of treatment with Secretol 80/80 versus Nexium 40 mg daily.

DETAILED DESCRIPTION:
We hypothesize that Secretol 80/80 daily will demonstrate better efficacy than Nexium 40 mg daily in healing erosive esophagitis(EE)and controlling gastroesophageal reflux disease(GERD)related symptoms after 3 weeks of treatment.In addition, Secretol 80/80 daily will have a faster effect on the aforementioned clinical parameters but a similar safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages 18-75
* EE Los Angeles grades C or D
* Heartburn and/or regurgitation at least 3 times a week during the 7 day run- in period prior to randomization.
* Able to read, understand, and complete study questionnaires and record
* Able to understand the study procedures and sign informed consent
* Able to comply with all study requirements

Exclusion Criteria:

* Subjects with Barrett's esophagus, non-erosive reflux disease,EE grades A or B, or peptic stricture on endoscopy
* Subjects with previous upper gastrointestinal surgery
* Subjects with clinically significant underlying comorbidity
* Helicobacter pylori positive
* Clinically significant GI bleed within the last 3 months
* Esophagitis not related to acid reflux
* Bleeding disorder
* Zollinger-Ellison, achalasia,esophageal varices, duodenal/gastric ulcer, upper gastrointestinal malignancy
* Women pregnant or lactating
* History of allergic reaction to any Proton Pump Inhibitor (PPI)
* Patients can't be treated concurrently with warfarin or other anticoagulants,salicylates,steroids,NSAIDS > 3 times/week
* Any medication dependant on gastric acid for optimal absorption

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Primary objective is to evaluate the relationship between healing and study drug allotment. | 3 weeks of treatment
  The primary objective is to evaluate the relationship between healing and study drug allotment. The variables to be used are erosive esophagitis healing status after 3 weeks of treatment as assessed by EGD (upper endoscopy) comparing to base line EGD.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Fass, MD, Principal Investigator — Southern Arizona VA Health Care System
Locations (1):
- Southern Arizona Veterans Health Care System, Tucson, Arizona, United States